CLINICAL TRIAL: NCT03524040
Title: Imaging of Pilosebaceous Units and Acne Lesions by Reflectance Confocal Microscopy and Optical Coherence Tomography
Brief Title: Imaging of Pilosebaceous Units and Acne Lesions by RCM and OCT Confocal Microscopy and Optical Coherence Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Collaborators: Sebacia, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, DMSc, PhD, MD, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-16042830
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Acne Vulgaris
Keywords: Selective Photothermolysis; Reflectance Confocal Microscopy; Optical Coherence Tomography; Pilosebaceous Unit; Gold Microparticles
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acne patients (Experimental): Application of gold microparticles to 2-3 facial areas
  Interventions: Device: SEB-250
- Heatlhy volunteers (Experimental): Application of gold microparticles to 2 facial areas
  Interventions: Device: SEB-250

INTERVENTIONS:
Device: SEB-250 — Gold microparticles (SEB-250) are massaged into 2 or 3 2x2 cm facial areas and exposed to 2 pulses from a diode laser

SUMMARY:
The purpose of the study was to investigate if reflectance confocal microscopy (RCM) and optical coherence tomography (OCT) could be used in combination to investigate the morphology of pilosebaceous units and acne lesions in healthy subjects and in acne patients.Furthermore, to investigate contrast effects, biodistribution and selective photothermolysis provided by gold microparticles and diode laser pulses, using RCM, OCT and histology.

ELIGIBILITY:
Inclusion Criteria:

All subjects

1. Healthy men and women
2. 18-45 years of age at baseline
3. Legally competent, able to give verbal and written consent
4. Communicate in Danish verbally as well as in writing
5. Women with negative pregnancy-test
6. Subject in good general health, is willing to participate and able to give informed consent, and can comply with protocol requirements.
7. Fitzpatrick skin phototype I-III

Acne skin

1. Subject with previous or prior clinical diagnosis of acne vulgaris, IGA score 1-4
2. Subjects with 1 - 75 inflammatory facial lesions on the cheek, forehead, and/or chin, with no more than 2 nodulocystic lesions (see Appendix II, table 4)
3. Each included patient with acne should represent at least 3 of 5 acne lesions
4. Subject with in good general health, willing to participate and able to give informed consent, and able to comply with protocol requirements

Exclusion Criteria:

1. Pregnant and lactating women
2. Subject with a known allergy to gold, or any other ingredient in the microparticle suspension
3. Individuals with skin diseases or skin lesions in the area of research interest will be excluded
4. Subject with tattoo in the treatment area which may interfere with or confound evaluation of the study
5. Subjects with severe acne (IGA 5) with imminent scarring potential, in the opinion of the investigator
6. Subject with a history of keloids which is deemed clinically relevant in the opinion of the investigator
7. Subject with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), or very severe acne requiring the continuation of systemic treatment during the study period.
8. Subject with active skin disease or excessive scarring that, in the opinion of the investigator, would impact the ability to administer the gold microparticles or use of OCT/RCM in the areas
9. Subject having used oral retionoid therapy such as isotretionoin within 3 months prior to baseline.
10. Subject having used topical retinoids, topical corticosteroids, topical antibiotics or combination therapy within 2 weeks of baseline
11. Subject having used over-the-counter topical products containing azelaic acid, benzoyl peroxide, and/or salicylic acid within 1 week of baseline
12. Subject having used light treatments including Intense Pulsed Light or other lasers, microdermabrasion or chemical peels in the treatment area within 3 weeks of baseline.
13. Subject who has received an investigational drug or was treated with an investigational device within 30 days prior to baseline.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Acne morphology | 1 year
  Qualitative assessment of acne lesions, pilosebaceous units and surrounding skin in RCM and OCT images
Gold microparticle biodistribution | 2 years
  Evaluation of gold microparticle biodistribution and contrast effects in RCM and OCT images

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided